CLINICAL TRIAL: NCT00943111
Title: A Phase 3, Randomized, Multi-Center, Multi-National, Open-Label, Active Comparator Study to Evaluate the Efficacy and Safety of Genz-112638 in Patients With Gaucher Disease Type 1 Who Have Reached Therapeutic Goals With Enzyme Replacement Therapy (ENCORE)
Brief Title: A Study of Eliglustat Tartrate (Genz-112638) in Patients With Gaucher Disease Who Have Reached Therapeutic Goals With Enzyme Replacement Therapy (ENCORE)
Acronym: ENCORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZGD02607; 2008-005223-28 (EudraCT Number); EFC12812 (Other: Sanofi)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Gaucher Disease, Type 1
Keywords: Gaucher disease,; Genz-112638,; beta-glucosidase,; acid ß-glucosidase,; glucocerebrosidase,; glucosylceramide,; D-glucosyl-N-acylsphingosine glucohydrolase,; substrate reduction therapy
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat; imiglucerase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational (Experimental): Eliglustat tartrate
  Interventions: Drug: Eliglustat tartrate
- Imiglucerase (Active Comparator)
  Interventions: Drug: Imiglucerase

INTERVENTIONS:
Drug: Eliglustat tartrate — Primary analysis period (PAP): Eliglustat tartrate capsule 50 milligram (mg) twice daily (BID) orally from Day 1 to Week 4 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 8, and then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to Week 52. Dose adjustments after Week 4 and Week 8 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations. If Genz-99067 trough plasma concentration was less than (<) 5 nanogram per milliliter [ng/mL] next higher dose was administered whereas if Genz-99067 trough plasma concentration was greater than or equal to (>=) 5 ng/mL same dose was continued. Pharmacokinetic (PK) assessment at Week 2 and 6 were used for dose adjustment after Week 4 and Week 8, respectively.
  Long-term treatment period (LTTP): Participants originally randomized to eliglustat in PAP continued to receive eliglustat dose, based on their Genz 99067 plasma trough concentration at Week 6.
  Other Names: Genz-112638
  Arms: Investigational
Drug: Imiglucerase — PAP: Imiglucerase intravenous infusion every other week (q2w) up to Week 52 in doses equivalent to participant's past ERT dose prior to any unanticipated treatment interruption, dose reduction, or regimen change.
  LTTP: Participants originally randomized to imiglucerase received eliglustat tartrate capsule 50 mg BID orally from Week 52+1 Day to Week 56 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 60, and then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to 5 years. The dose adjustments after Week 56 and Week 60 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations. If Genz-99067 trough plasma concentration was <5 ng/mL the next higher dose was administered whereas if the Genz-99067 trough plasma concentration was >=5 ng/mL the same dose was continued. The PK assessment at Week 54 and Week 58 were used for dose adjustment after Week 56 and Week 60, respectively.
  Other Names: Cerezyme®
  Arms: Imiglucerase

SUMMARY:
This Phase 3 study was designed to confirm the efficacy and safety of eliglustat tartrate (Genz-112638) in participants with Gaucher disease type 1 who had reached therapeutic goals with enzyme replacement therapy (ERT).

DETAILED DESCRIPTION:
Gaucher disease is characterized by lysosomal accumulation of glucosylceramide due to impaired glucosylceramide hydrolysis. Gaucher disease type 1, which is the most common form, accounts for greater than (>) 90% of cases and does not involve the central nervous system (CNS). Typical manifestations of Gaucher disease type 1 include splenomegaly, hepatomegaly, thrombocytopenia, anemia, bone disease, and decreased quality of life. The disease manifestations are caused by the accumulation of glucosylceramide (storage material) in macrophages (called Gaucher cells) which have infiltrated the spleen and liver as well as other tissues.

Eliglustat tartrate is a small molecule drug developed as an oral therapy which acts to specifically inhibit production of this storage material in Gaucher cells.

This study was designed to determine the efficacy, safety, and PK of eliglustat tartrate in adult participants with Gaucher disease type 1 who had been stabilized on ERT.

ELIGIBILITY:
Inclusion Criteria:

* The participant (and/or their parent/legal guardian) was willing and able to provide signed informed consent prior to any study-related procedures to be performed
* The participant was at least 18 years old at the time of randomization
* The participant had a confirmed diagnosis of Gaucher disease type 1
* The participant had received treatment with ERT for at least 3 years. Within the 9 months prior to randomization, the participant had received a total monthly dose of 30 to 130 Units/kilogram for at least 6 months
* The participant had reached Gaucher disease therapeutic goals prior to randomization
* Female participants of childbearing potential must have had a documented negative pregnancy test prior to dosing. In addition, all female participants of childbearing potential must use a medically accepted form of contraception throughout the study

Exclusion Criteria:

* The participant had a partial or total splenectomy within 3 years prior to randomization
* The participant had received substrate reduction therapies for Gaucher disease within 6 months prior to randomization
* The participant had Gaucher disease type 2 or 3 or was suspected of having Gaucher disease type 3
* The participant had any clinically significant disease, other than Gaucher disease, including cardiovascular, renal, hepatic, gastrointestinal (GI), pulmonary, neurologic, endocrine, metabolic (e.g. hypokalemia, hypomagnesemia), or psychiatric disease, other medical conditions, or serious intercurrent illnesses that may confound the study results or, in the opinion of the Investigator, may preclude participation in the study
* The participant had tested positive for the human immunodeficiency virus (HIV) antibody, Hepatitis C antibody, or Hepatitis B surface antigen
* The participant had received an investigational product within 30 days prior to randomization
* The participant was pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (34):
- United States (17):
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - UCSF MS Center, San Francisco, California
  - University of Colorado Health Science Center - Aurora, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Northwest Oncology Hematology Associates PA, Coral Springs, Florida
  - Emory University Medical Genetics, Decatur, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albany Medical Center, Albany, New York
  - North Shore University Medical Center, Manhasset, New York
  - Mount Sinai School of Medicine, New York, New York
  - New York University School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - O and O Alpan LLC, Springfield, Virginia
- Argentina (2):
  - Hospital General de Agudos J.M Ramos Mejia, Buenos Aires
  - Hospital General de Ninos Dr. Ricardo Gutierrez, Buenos Aires
- Royal Perth Hospital, Perth, WA, Australia
- Brazil (3):
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba
  - Instituto de Estadual de Hematologia Arthur de Siqueria Cavalcanti, Rio de Janeiro
  - IGEIM, São Paulo
- Mount Sinai Hospital and the Samuel Lunenfeld Research Institute, Toronto Ontario, Canada
- Abou El Reesh Children's University Hospital (El Mounira), Faculty of Medicine (Kasr Al-Aini), Cairo University Hospitals, El Mounira, Cairo, Egypt, Cairo, Egypt
- Hôpital Beaujon, Clichy, France
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - Asklepios Klinik St. Georg, Hamburg
  - Katholische Kliniken Oberhausen gem. GmbH, Oberhausen
- Italy (2):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedialiero-Universitaria S. Maria Della Misericordia, Udine
- Hematology Research Center of Ministry of Healthcare of the Russian Federation, Moscow, Russia
- Hospital University Miguel Servet, Zaragoza, Spain
- Cambridge University Hosptials, Addenbrookes Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Lukina E, Watman N, Arreguin EA, Banikazemi M, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Rosenthal DI, Kaper M, Singh T, Puga AC, Bonate PL, Peterschmitt MJ. A phase 2 study of eliglustat tartrate (Genz-112638), an oral substrate reduction therapy for Gaucher disease type 1. Blood. 2010 Aug 12;116(6):893-9. doi: 10.1182/blood-2010-03-273151. Epub 2010 May 3. PMID 20439622
- [Background] Lukina E, Watman N, Arreguin EA, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Kamath RS, Rosenthal DI, Kaper M, Singh T, Puga AC, Peterschmitt MJ. Improvement in hematological, visceral, and skeletal manifestations of Gaucher disease type 1 with oral eliglustat tartrate (Genz-112638) treatment: 2-year results of a phase 2 study. Blood. 2010 Nov 18;116(20):4095-8. doi: 10.1182/blood-2010-06-293902. Epub 2010 Aug 16. PMID 20713962
- [Background] McEachern KA, Fung J, Komarnitsky S, Siegel CS, Chuang WL, Hutto E, Shayman JA, Grabowski GA, Aerts JM, Cheng SH, Copeland DP, Marshall J. A specific and potent inhibitor of glucosylceramide synthase for substrate inhibition therapy of Gaucher disease. Mol Genet Metab. 2007 Jul;91(3):259-67. doi: 10.1016/j.ymgme.2007.04.001. Epub 2007 May 16. PMID 17509920
- [Background] Kamath RS, Lukina E, Watman N, Dragosky M, Pastores GM, Arreguin EA, Rosenbaum H, Zimran A, Aguzzi R, Puga AC, Norfleet AM, Peterschmitt MJ, Rosenthal DI. Skeletal improvement in patients with Gaucher disease type 1: a phase 2 trial of oral eliglustat. Skeletal Radiol. 2014 Oct;43(10):1353-60. doi: 10.1007/s00256-014-1891-9. Epub 2014 May 10. PMID 24816856
- [Background] Lukina E, Watman N, Dragosky M, Pastores GM, Arreguin EA, Rosenbaum H, Zimran A, Angell J, Ross L, Puga AC, Peterschmitt JM. Eliglustat, an investigational oral therapy for Gaucher disease type 1: Phase 2 trial results after 4 years of treatment. Blood Cells Mol Dis. 2014 Dec;53(4):274-6. doi: 10.1016/j.bcmd.2014.04.002. Epub 2014 May 15. PMID 24835462
- [Derived] Cox TM, Drelichman G, Cravo R, Balwani M, Burrow TA, Martins AM, Lukina E, Rosenbloom B, Goker-Alpan O, Watman N, El-Beshlawy A, Kishnani PS, Pedroso ML, Gaemers SJM, Tayag R, Peterschmitt MJ. Eliglustat maintains long-term clinical stability in patients with Gaucher disease type 1 stabilized on enzyme therapy. Blood. 2017 Apr 27;129(17):2375-2383. doi: 10.1182/blood-2016-12-758409. Epub 2017 Feb 6. PMID 28167660
- [Derived] Cox TM, Drelichman G, Cravo R, Balwani M, Burrow TA, Martins AM, Lukina E, Rosenbloom B, Ross L, Angell J, Puga AC. Eliglustat compared with imiglucerase in patients with Gaucher's disease type 1 stabilised on enzyme replacement therapy: a phase 3, randomised, open-label, non-inferiority trial. Lancet. 2015 Jun 13;385(9985):2355-62. doi: 10.1016/S0140-6736(14)61841-9. Epub 2015 Mar 26. PMID 25819691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 209 participants were screened, of which 46 participants were screen failure and 3 participants withdrew prior to randomization. A total of 160 participants were enrolled in this study.
Pre-assignment Details: All enrolled participants received eliglustat or imiglucerase in 52 week primary analysis period (PAP). After 52-weeks PAP, all participants who remained on-study, received eliglustat in the long-term treatment period (LTTP) for up to 5 years.
Groups:
- Eliglustat: PAP: Eliglustat tartrate (Genz-112638) capsule 50 milligram (mg) twice daily (BID) orally from Day 1 to Week 4 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 8, and then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to Week 52. The dose adjustments after Week 4 and Week 8 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations. If Genz-99067 trough plasma concentration was less than [<] 5 nanogram per milliliter [ng/mL] the next higher dose was administered whereas if the Genz-99067 trough plasma concentration was greater than or equal to [>=] 5 ng/mL the same dose was continued. The pharmacokinetic (PK) assessment at Week 2 and Week 6 were used for dose adjustment after Week 4 and Week 8, respectively.
- Imiglucerase: PAP: Imiglucerase (Cerezyme®) intravenous infusion every other week (q2w) up to Week 52 in doses equivalent to participant's past enzyme replacement therapy (ERT) dose prior to any unanticipated treatment interruption, dose reduction, or regimen change.
- Eliglustat: LTTP: Participants from both the arms of PAP who completed PAP were included in this arm of LTTP.
  Participants originally randomized to eliglustat in PAP continued to receive eliglustat dose, based on their Genz 99067 plasma trough concentration at Week 6.
  Participants originally randomized to imiglucerase received eliglustat tartrate capsule 50 mg BID orally from Week 52+1 Day to Week 56 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 60, and then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to 5 years. The dose adjustments after Week 56 and Week 60 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations. If Genz-99067 trough plasma concentration was <5 ng/mL next higher dose was administered whereas if the Genz-99067 trough plasma concentration was >=5 ng/mL the same dose was continued. PK assessment at Week 54 and Week 58 were used for dose adjustment after Week 56 and Week 60, respectively.
Period: 52-Weeks Primary Analysis Period
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP | Eliglustat: LTTP
Started | 106 | 54 | 0
Treated | 106 | 53 | 0
Completed | 104 | 52 | 0
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 1 | 0
Period: 5 Years Long-term Treatment Period
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP | Eliglustat: LTTP
Started | 0 | 0 | 152 (Participants from both the arms of PAP who completed PAP and remained on-study)
Completed | 0 | 0 | 77
Not Completed | 0 | 0 | 75
Not completed — Transition to commercial eliglustat | 0 | 0 | 51
Not completed — Adverse Event | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 8
Not completed — Pregnancy | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other than specified above | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) for PAP: included all participants who signed informed consent and received at least 1 dose of study drug (Imiglucerase or eliglustat).
Groups:
- Eliglustat: PAP: Eliglustat tartrate 50 mg capsule BID orally from Day 1 to Week 4, followed by eliglustat tartrate 50, 100 or 150 mg capsule BID orally up to Week 52.
- Imiglucerase: PAP: Imiglucerase intravenous infusion q2w up to Week 52 in doses equivalent to participant's past ERT dose prior to any unanticipated treatment interruption, dose reduction, or regimen change.
- Total: Total of all reporting groups
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP | Total
Number analyzed (Participants) | 106 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (14.17) | 37.5 (14.92) | 37.5 (14.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 28 | 87
  Male | 47 | 25 | 72
Race/Ethnicity, Customized [Number; unit: participants]
  Race: White | 98 | 48 | 146
  Race: Black or African American | 6 | 4 | 10
  Race: Asian | 1 | 1 | 2
  Race: White/American Indian | 1 | 0 | 1
  Ethnicity: Hispanic or Latino | 42 | 19 | 61
  Ethnicity: Not Hispanic or Latino | 64 | 34 | 98
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated as ([weight in kg] divided by [height in cm multiplied by 0.01]^2).
  kilogram per square meter (kg/m^2) | 25.2 (5.24) | 24.5 (4.51) | 24.9 (5.01)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 70.8 (16.82) | 67.8 (14.44) | 69.8 (16.08)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 167.6 (9.92) | 166.2 (9.56) | 167.1 (9.79)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Remained Stable for 52 Weeks During the Primary Analysis Period
Description: For a participant to be classified as stable, the participant must have remained stable in hematological parameters (hemoglobin levels and platelet counts) and organ volumes (spleen, when applicable, and liver volumes in multiples of normal [MN]). Stable hematological parameters were defined as hemoglobin level did not decrease more than (>) 1.5 gram per deciliter (g/dL) from baseline and platelet count did not decrease >25% from baseline. Stable organ volumes were defined as spleen volume (in MN) did not increase >25% from baseline, if applicable, and liver volume (in MN) did not increase >20% from baseline.
Time Frame: Baseline up to Week 52
Population: Per protocol population for PAP included participants who were at least 80% compliant with treatment during PAP, had no major protocol deviations, and did not exhibit hematological decline as a result of medically determined etiologies other than Gaucher disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 99 | 47
percentage of participants | 84.8 [76.2 to 91.3] | 93.6 [82.5 to 98.7]
Statistical Analysis 1: Comparison: Eliglustat: PAP vs Imiglucerase: PAP; Test type: Non-Inferiority or Equivalence — The sample size for study was based on expected stability rates of 95% for the Imiglucerase group and 85% for the Eliglustat group, power of 85%, a one-sided significance level of 0.025, a non-inferiority margin of 25%, and a 20% non-evaluable/drop-out rate. Eliglustat was declared non-inferior to Imiglucerase if the lower-bound of the 95% confidence interval for the difference was within the non-inferiority margin of 25%; Difference in Percentage Stable = -8.8, 95% CI 2-sided [-17.6 to 4.2]

2. Primary Outcome: Percentage of Participants Who Remained Stable Annually for 4 Years During the LTTP
Description: For a participant to be classified as stable, the participant must have remained stable in hematological parameters (hemoglobin levels and platelet counts) and organ volumes (spleen, when applicable, and liver volumes in MN). Stable hematological parameters were defined as hemoglobin level did not decrease >1.5 g/dL from baseline and platelet count did not decrease >25% from baseline. Stable organ volumes were defined as spleen volume (in MN) did not increase >25% from baseline, if applicable, and liver volume did not increase >20% from baseline.
Time Frame: Week 52 up to week 208
Population: FAS population for LTTP: included all participants who received at least 1 dose of eliglustat in the extension study period. Number of participants analyzed=participants at risk at specified time-points. Here 'n' signifies number of participants with available data for specified time-points.
Measure: Number; unit: percentage of participants
Groups:
- Eliglustat: LTTP: Participants from both the arms of PAP who completed PAP were included in this arm of LTTP.
  Participants originally randomized to eliglustat in PAP continued to receive eliglustat dose, based on their Genz 99067 plasma trough concentration at Week 6.
  Participants originally randomized to imiglucerase received eliglustat tartrate capsule 50 mg BID orally from Week 52+1 Day to Week 56 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 60, and then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to 5 years. The dose adjustments after Week 56 and Week 60 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations.
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 152
percentage of participants
  Year 1 (n=127) | 83.6
  Year 2 (n= 115) | 75.65
  Year 3 (n= 92) | 60.53
  Year 4 (n= 41) | 26.97

3. Secondary Outcome: Total T-Scores for Bone Mineral Density
Description: Images of the spine and bilateral femur were obtained by dual energy X-Ray absorptiometry (DXA) to determine T-score for each bone area and total bone mineral density. T-score compares participant's bone density with that of healthy young participant. The T-score bone density categories are: normal (score greater than [>]-1), osteopenia (score -2.5 to less than or equal to [<=] -1), and osteoporosis (score <= -2.5).
Time Frame: Baseline
Population: Per protocol population for PAP. Number of participants analyzed = participants with baseline T-score assessment. Here, 'n' signifies participants with baseline T-score assessment for specified bone area.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 81 | 38
T-score
  Lumbar Spine T-Score (n=81, 38) | -0.56 (1.309) | -0.33 (1.169)
  Femur T-Score (n=80, 37) | -0.11 (1.080) | -0.47 (1.293)

4. Secondary Outcome: Absolute Change From Baseline in Total T-Scores for Bone Mineral Density at Week 52
Description: Images of the spine and bilateral femur were obtained by DXA to determine T-score for each bone area and total bone mineral density. T-score compares participant's bone density with that of healthy young participant. The T-score bone density categories are: normal (score >-1), osteopenia (score -2.5 to <=-1), and osteoporosis (score <= -2.5). Absolute change = T-score at Week 52 minus T-score at baseline.
Time Frame: Baseline, Week 52
Population: Per protocol population for PAP. Number of participants analyzed = participants with both baseline and Week 52 T-score assessment. Here, 'n' signifies participants with both baseline and Week 52 T-score assessment for specified bone area. Eliglustat participants switching to imiglucerase were excluded.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 81 | 38
T-score
  Change in Lumbar Spine T-Score (n=81, 38) | 0.04 (0.03) | 0.03 (0.05)
  Change in Femur T-Score (n=80, 37) | 0.00 (0.02) | -0.03 (0.03)

5. Secondary Outcome: Total Z-Scores for Bone Mineral Density
Description: Images of the spine and bilateral femur were obtained by DXA to determine Z-score for each bone area and total bone mineral density. The Z-score bone density categories are: normal (score >-2) and below normal (score <=-2).
Time Frame: Baseline
Population: Per protocol population for PAP. Number of participants analyzed = participants with baseline Z-score assessment. Here, 'n' signifies participants with baseline Z-score assessment for specified bone area.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 94 | 45
Z-score
  Lumbar Spine Z-Score (n=94, 45) | -0.35 (1.260) | -0.14 (1.108)
  Femur Z-Score (n=93, 44) | 0.09 (1.020) | -0.18 (1.122)

6. Secondary Outcome: Absolute Change From Baseline in Total Z-Scores for Bone Mineral Density at Week 52
Description: Images of the spine and bilateral femur were obtained by DXA to determine Z-score for each bone area and total bone mineral density. The Z-score bone density categories are: normal (score >-2) and below normal (score <=-2). Absolute change = Z-score at Week 52 minus Z-score at baseline.
Time Frame: Baseline, Week 52
Population: Per protocol population for PAP. Number of participants analyzed = participants with both baseline and Week 52 Z-score assessment. Here, 'n' signifies participants with both baseline and Week 52 Z-score assessment for specified bone area. Eliglustat participants switching to imiglucerase were excluded.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 94 | 45
Z-score
  Change in Lumbar Spine Z-Score (n=94, 45) | 0.06 (0.03) | 0.06 (0.04)
  Change in Femur Z-Score (n=93, 44) | 0.03 (0.02) | 0.02 (0.02)

7. Secondary Outcome: Hemoglobin Level
Time Frame: Baseline
Population: Per protocol population for PAP. Number of participants analyzed = participants with baseline hemoglobin assessment.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 98 | 47
gram per deciliter (g/dL) | 13.592 (1.2467) | 13.797 (1.2234)

8. Secondary Outcome: Absolute Change From Baseline in Hemoglobin Levels at Week 52
Description: Absolute change = hemoglobin level at Week 52 minus hemoglobin level at baseline.
Time Frame: Baseline, Week 52
Population: Per protocol population for PAP. Number of participants analyzed = participants with both baseline and Week 52 hemoglobin assessment. Eliglustat participants switching to imiglucerase were excluded.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 98 | 47
g/dL | -0.22 (0.07) | 0.05 (0.10)

9. Secondary Outcome: Percent Change From Baseline in Platelet Counts at Week 52
Description: Percent change in platelet counts = ([platelet count at Week 52 minus platelet count at baseline] divided by [platelet count at baseline]) multiplied by 100.
Time Frame: Baseline, Week 52
Population: Per protocol population for PAP. Number of participants analyzed = participants with both baseline and Week 52 platelet assessment. Eliglustat participants switching to imiglucerase were excluded.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 98 | 47
percent change | 3.93 (1.71) | 2.63 (2.47)

10. Secondary Outcome: Percent Change From Baseline in Spleen Volume (MN) at Week 52
Description: Percent change in spleen volume = ([spleen volume at Week 52 minus spleen volume at baseline] divided by [spleen volume at baseline]) multiplied by 100, where all volumes are in MN.
Time Frame: Baseline, Week 52
Population: Per protocol population for PAP. Number of participants analyzed = participants with both baseline and Week 52 spleen volume assessment. Eliglustat participants switching to imiglucerase were excluded.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 70 | 39
percent change | -6.05 (1.57) | -3.22 (2.13)

11. Secondary Outcome: Percent Change From Baseline in Liver Volume (in MN) at Week 52
Description: Percent change in liver volume = ([liver volume at Week 52 minus liver volume at baseline] divided by [liver volume at baseline]) multiplied by 100, where all volumes are in multiples of normal.
Time Frame: Baseline, Week 52
Population: Per protocol population for PAP. Number of participants analyzed = participants with both baseline and Week 52 liver volume assessment. Eliglustat participants switching to imiglucerase were excluded.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Eliglustat: PAP | Imiglucerase: PAP
Number analyzed (Participants) | 98 | 47
percent change | 1.99 (0.94) | 3.13 (1.36)

12. Secondary Outcome: Absolute Change From Baseline in Total T-Scores for Bone Mineral Density at Week 208
Description: Images of the spine and bilateral femur were obtained by DXA to determine T-score for each bone area and total bone mineral density. T-score compares participant's bone density with that of healthy young participant. The T-score bone density categories are: normal (score >-1), osteopenia (score -2.5 to <=-1), and osteoporosis (score <= -2.5). Absolute change = T-score at Week 208 minus T-score at baseline.
Time Frame: Baseline, Week 208
Population: Number of participants analyzed = participants with both baseline and Week 208 T-score assessment.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 36
T-Score
  Total Spine | 0.22 (0.405)
  Total Femur | -0.03 (0.345)

13. Secondary Outcome: Absolute Change From Baseline in Total Z-Scores for Bone Mineral Density at Week 208
Description: Images of the spine and bilateral femur were obtained by DXA to determine Z-score for each bone area and total bone mineral density. The Z-score bone density categories are: normal (score >-2) and below normal (score <=-2). Absolute change = Z-score at Week 208 minus Z-score at baseline.
Time Frame: Baseline, Week 208
Population: FAS population for LTTP. Number of participants analyzed = participants with both baseline and Week 208 Z-score assessment. Here, 'n' signifies participants with both baseline and Week 208 Z-score assessment for specified bone area.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 42
Z-score
  Total Spine | 0.29 (0.358)
  Total Femur | 0.03 (0.381)

14. Secondary Outcome: Absolute Change From Baseline in Hemoglobin Levels at Week 208
Description: Absolute change = hemoglobin level at Week 208 minus hemoglobin level at baseline.
Time Frame: Baseline, Week 208
Population: FAS population for LTTP. Number of participants analyzed = participants with both baseline and Week 208 hemoglobin assessment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 45
g/dL | 0.297 (0.7472)

15. Secondary Outcome: Percent Change From Baseline in Platelet Counts at Week 208
Description: Percent change in platelet counts = ([platelet count at Week 208 minus platelet count at baseline] divided by [platelet count at baseline]) multiplied by 100.
Time Frame: Baseline, Week 208
Population: FAS population for LTTP. Number of participants analyzed = participants with both baseline and Week 208 platelet assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 45
percent change | 6.990 (20.4382)

16. Secondary Outcome: Percent Change From Baseline in Spleen Volume (in MN) at Week 208
Description: Percent change in spleen volume = ([spleen volume at Week 208 minus spleen volume at baseline] divided by [spleen volume at baseline]) multiplied by 100, where all volumes are in MN.
Time Frame: Baseline, Week 208
Population: FAS population for LTTP. Number of participants analyzed = participants with both baseline and Week 208 spleen volume assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 33
percent change | -14.768 (17.9435)

17. Secondary Outcome: Percent Change From Baseline in Liver Volume (in MN) at Week 208
Description: Percent change in liver volume = ([liver volume at Week 208 minus liver volume at baseline] divided by [liver volume at baseline]) multiplied by 100, where all volumes are in multiples of normal.
Time Frame: Baseline, Week 208
Population: FAS population for LTTP. Number of participants analyzed = participants with both baseline and Week 208 liver volume assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat: LTTP
Number analyzed (Participants) | 46
percent change | -2.345 (12.8795)

ADVERSE EVENTS:
Time Frame: From signature of informed consent up to 30-37 days after the last dose of treatment (last dose = up to Week 104)
Description: Safety set included all participants who received at least 1 dose of study drug (Eliglustat or Imiglucerase). In the event a single participant experienced both serious and non-serious forms of same adverse events (AE), individual was included in numerator (number of participants affected) of each AE table.
Groups:
- Eliglustat: PAP: Eliglustat tartrate 50 mg capsule BID orally from Day 1 to Week 4, followed by eliglustat tartrate 50, 100 or 150 mg capsule BID orally up to Week 52. Dose adjustments after Week 4 and Week 8 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations. LTTP: Participants originally randomized to eliglustat in PAP continued to receive eliglustat dose, based on their Genz 99067 plasma trough concentration at Week 6.
- Imiglucerase: PAP: Imiglucerase (Cerezyme®) intravenous infusion q2w up to Week 52 in doses equivalent to participant's past ERT dose prior to any unanticipated treatment interruption, dose reduction, or regimen change. LTTP: Participants originally randomized to imiglucerase received eliglustat tartrate capsule 50 mg BID orally from Week 52+1 Day to Week 56 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 60, and then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to 5 years. The dose adjustments after Week 56 and Week 60 were based on Genz-99067 (active moiety of eliglustat tartrate in plasma) trough plasma concentrations.
Arm/Group | Eliglustat | Imiglucerase
Serious Adverse Events (participants affected / at risk) | 18/106 | 7/53
Other Adverse Events (participants affected / at risk) | 91/106 | 38/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat (N=106) | Imiglucerase (N=53)
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mammoplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat (N=106) | Imiglucerase (N=53)
Palpitations (Cardiac disorders) | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 6
Abdominal pain lower (Gastrointestinal disorders) | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 26 | 3
Constipation (Gastrointestinal disorders) | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 20 | 2
Dyspepsia (Gastrointestinal disorders) | 15 | 4
Gastritis (Gastrointestinal disorders) | 6 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 2
Nausea (Gastrointestinal disorders) | 18 | 7
Toothache (Gastrointestinal disorders) | 7 | 3
Vomiting (Gastrointestinal disorders) | 10 | 0
Asthenia (General disorders) | 10 | 1
Chest pain (General disorders) | 9 | 1
Fatigue (General disorders) | 20 | 7
Pain (General disorders) | 6 | 3
Peripheral swelling (General disorders) | 6 | 1
Pyrexia (General disorders) | 2 | 3
Hepatomegaly (Hepatobiliary disorders) | 5 | 3
Bronchitis (Infections and infestations) | 8 | 2
Gastroenteritis (Infections and infestations) | 11 | 2
Influenza (Infections and infestations) | 20 | 6
Nasopharyngitis (Infections and infestations) | 28 | 10
Sinusitis (Infections and infestations) | 20 | 3
Upper respiratory tract infection (Infections and infestations) | 21 | 7
Urinary tract infection (Infections and infestations) | 16 | 3
Contusion (Injury, poisoning and procedural complications) | 7 | 2
Laceration (Injury, poisoning and procedural complications) | 7 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 8 | 0
Limb injury (Injury, poisoning and procedural complications) | 6 | 0
Blood creatine phosphokinase increased (Investigations) | 16 | 3
Mean cell volume abnormal (Investigations) | 0 | 3
Nerve conduction studies abnormal (Investigations) | 7 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 5
Dizziness (Nervous system disorders) | 18 | 4
Headache (Nervous system disorders) | 26 | 9
Hypoaesthesia (Nervous system disorders) | 6 | 1
Paraesthesia (Nervous system disorders) | 7 | 1
Anxiety (Psychiatric disorders) | 10 | 1
Depression (Psychiatric disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Hypertension (Vascular disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.